CLINICAL TRIAL: NCT00904423
Title: A Phase I/II Randomized, Double-blind, Controlled Study to Evaluate Efficacy and Safety of Vitamin D on Bone Mineral Density and Markers of Bone Resorption in Aromatase Inhibitor-induced Bone Loss in Women With Breast Cancer.
Brief Title: Ph I/II of Vitamin D on Bone Mineral Density & Markers of Bone Resorption
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low accrual
Sponsor: Mark Pegram (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor-Investigator, Mark Pegram, Susy Yuan-Huey Hung Professor, Stanford University
Organization: Stanford University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB-15005; SU-09232008-1302 (Other: Stanford University); BRSADJ0014 (Other: OnCore)
Record Dates: First submitted 2009-05-13; First posted 2009-05-19 (Estimated); Results first posted 2017-02-14 (Actual); Last update posted 2017-02-14 (Actual); Status verified 2016-12

CONDITIONS: Breast Cancer; Bone Diseases
MeSH Terms: conditions — Breast Neoplasms; Bone Diseases | interventions — Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Vitamin D (Experimental)
  Interventions: Drug: Vitamin D

INTERVENTIONS:
Drug: Vitamin D — up to 2400 mg; oral tablet
  Other Names: Vital nutrients

SUMMARY:
Aromatase inhibitors are potent suppressors of breast cancer growth, but side effects include bone loss, fractures, arthralgias and myalgias. We hypothesize vitamin D administration might be beneficial in treating these symptoms and to protect bone.

ELIGIBILITY:
Inclusion Criteria:

3.1.1 All postmenopausal women with histology-confirmed invasive primary breast cancer, who have completed primary surgical or radiotherapy (XRT) with or without adjuvant chemotherapy and are candidates to receive adjuvant therapy with aromatase inhibitors will be screened for eligibility. Postmenopausal is defined as satisfying one or more of the following criteria: having had bilateral oophorectomy; aged more than 60 years; or aged 55-59 years with an intact uterus and amenorrheic for at least 12 months; or if amenorrheic for less than 12 months (after receiving hysterectomy, hormone therapy or chemotherapy).

3.1.2 At the time of study enrollment, participants will have completed primary surgical or XRT with or without adjuvant chemotherapy. Chemotherapy will be completed at least 28 days prior to enrollment.

3.1.4 Participants will be women between 18-85 years of age. Women and minorities will be actively recruited. Though breast cancer extremely rarely occurs in children and men, this study will only recruit adult females.

3.1.5 Participants will have a life expectancy of at least 5 years.

3.1.6 Participants will have Eastern Clinical Oncology Group (ECOG) performance status 0-2.

3.1.7 Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

3.2.1 Medications affecting bone metabolism (bisphosphonates, anticonvulsants, chronic heparin therapy, chronic glucocorticoid use > 5 mg/day prednisone or equivalent, teriparatide).

3.2.2 Use of any investigational drug within past 90 days.

3.2.3 Metastatic breast cancer. High risk for osteoporosis/fractures (BMD < -2.0, history of non-traumatic fracture). Hyperparathyroidism Hypercalcemia Hypercalciuria (fasting spot urine calcium/creatinine ratio >0.20) History of renal stones Renal failure with creatinine over 2.0

3.2.4 Considering that vitamin D3 is produced by the human body, allergy to vitamin D3 is not expected to develop. Subjects with known history of allergic reaction to compounds used to manufacture capsules (rice powder) will be excluded form this study.

3.2.5 Recent history of excessive alcohol or drug use.

3.2.6 As this study will recruit post-menopausal patients, thus pregnant or nursing patients are not part of this investigation.

3.2.8 This study is designed to study women after completing primary therapy for breast cancer. Survivors of previous cancers and HIV-positive subjects will not be excluded.

Ages: 18 Years to 85 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2009-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eva Balint, Principal Investigator — Stanford University; Robert W Carlson, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Vitamin D
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Vitamin D
Number analyzed (Participants) | 8
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 8
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 3
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 5
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Spine Bone Mineral Density T Score Change Over One Year
Time Frame: 1 year
Population: Data are not accessible.
Arm/Group | Vitamin D
Number analyzed (Participants) | 0

2. Secondary Outcome: Change in Hip Bone Mineral Density (BMD) T-score
Time Frame: one year
Population: Data are not accessible.
Arm/Group | Vitamin D
Number analyzed (Participants) | 0

3. Secondary Outcome: Bone Turnover Markers
Time Frame: months 4 and 12
Population: Data are not accessible.
Arm/Group | Vitamin D
Number analyzed (Participants) | 0

4. Secondary Outcome: Arthralgias and Myalgias
Time Frame: every 4 months
Population: Data are not accessible.
Arm/Group | Vitamin D
Number analyzed (Participants) | 0

5. Secondary Outcome: Serum Calcium and Fasting Spot Urine Calcium/Creatinine Ratio
Time Frame: every 4 months
Population: Data are not accessible.
Arm/Group | Vitamin D
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse event data are not accessible.
Arm/Group | Vitamin D
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 0/8

LIMITATIONS AND CAVEATS:
Early termination secondary to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No